CLINICAL TRIAL: NCT04987346
Title: Normative Database for Gait Analyses and Balance on the GRAIL at the University Hospital of Ghent.
Brief Title: Normative Database for Gait Analysis on the GRAIL UZ Gent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B670201942108
Record Dates: First submitted 2021-07-05; First posted 2021-08-03 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Gait
Keywords: Gait analysis; Control group; Healthy; Reference data; Kinematics; Kinetics; EMG; Dual-tasking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treadmill walking (Experimental): Participants will be asked to walk at different gait velocities for 1 minute. The treadmill speed will be increased incrementally at 0.1m/s intervals until just before running.
  Interventions: Other: Walking on an instrumented treadmill; Other: Walking on an instrumented treadmill while dual-tasking

INTERVENTIONS:
Other: Walking on an instrumented treadmill — Participants will be asked to walk at different gait velocities for 1 minute. The treadmill speed will be increased incrementally at 0.1m/s intervals until just before running.
Other: Walking on an instrumented treadmill while dual-tasking — Participants aged between 6 and 17 years will be asked to walk at comfortable walking speed while playing either a cognitive (Stroop Color and Word Test) or motor (requiring arm swing) game.

SUMMARY:
The aim of this study is to collect a large set of norm/control data on an instrumented treadmill (the Gait Real-time Analysis Interactive Lab - GRAIL) at the university hospital of Ghent for the purpose of clinical studies as well as for clinical interpretation.

We hypothesize that this norm/control data will provide reference data of the normal gait patterns in the healthy population such that we can then use it to identify gait abnormalities in populations with pathology.

The following data will be collected on the GRAIL while subjects walk at different gait speeds: 3D kinematics, kinetics, and EMG.

Additionally, 3D kinematics, kinetics, and EMG data will be collected when performing either a cognitive (Stroop Color and Word Test) or motor (requiring arm swing) dual-task while walking at comfortable walking speed.

ELIGIBILITY:
Inclusion Criteria:

- Healthy participants

Exclusion Criteria:

* They suffer from neurological disorder
* Have balance problems
* Take medications that affect gait and balance
* Have undergone surgical procedures on the lower limbs in the past
* Experience pain in their lower limbs or back at the time of test taking.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Kinematics | single point assessment in 1 day
  3D kinematics of lower and upper limb joints while walking (degrees)
Kinetics | single point assessment in 1 day
  3D kinetics of lower limb joints while walking (Nm)
EMG | single point assessment in 1 day
  Muscle activity of 32 lower and upper limb muscles (micorvolts)
EMG synergies | single point assessment in 1 day
  Synergy analysis will be carried using the EMG data (variance accounted for -VAF)
Spatiotemporal parameters | single point assessment in 1 day
  Spatial parameters (m)
Spatiotemporal parameters | single point assessment in 1 day
  Temporal parameters (s)
Spatiotemporal parameters | single point assessment in 1 day
  Walking velocity (m/s)

SECONDARY OUTCOMES:
Gait deviation index | single point assessment in 1 day
  Based on kinematics, the lower-limb gait deviations will be calculated (degrees)
Game result (cognitive task) | single point assessment in 1 day
  Score (% correct)
Game result (motor task) | single point assessment in 1 day
  Score (% correct)

OTHER OUTCOMES:
Demographic data | single point assessment in 1 day
  Gender, age
height (cm) | single point assessment in 1 day
  anthropometric data
weight | single point assessment in 1 day
  anthropometric data
segment lengths (cm) | single point assessment in 1 day
  anthropometric data
M-ABC-2 | single point assessment in 1 day
  Standardized tool to indentify motor functioning in children
Developmental Coordination Disorder Questionnaire (DCDQ) | single point assessment in 1 day
  Brief parent questionnaire to screen for coordination disorders in children

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No